CLINICAL TRIAL: NCT01135173
Title: Pilot Test of a Cessation Intervention for Waterpipe Smokers
Brief Title: Waterpipe Cessation Intervention Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Kenneth D. Ward, PhD, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H06-100-03
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation, Waterpipe
MeSH Terms: conditions — Smoking Cessation; Water Pipe Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Motivational and educational intervention, delivered by a trained physician from the SCTS plus written self-help materials.
  Interventions: Behavioral: Waterpipe smoking cessation
- Arm B (Experimental): Behavioral counseling intervention conducted by a trained physician at the SCTS cessation clinic. Subjects complete "homework" before the session to facilitate this process. Subjects are asked to identify high-risk situations and difficulties in previous cessation attempts and are walked through a series of suggestions in the event of a slip. Three brief (approximately 10 minute) phone calls are provided to subjects during the 90 day follow-up period. These calls are used to identify early relapse, encourage participants, and provide support. In addition, they are used to review materials and information provided during the sessions.
  Interventions: Behavioral: Waterpipe smoking cessation

INTERVENTIONS:
Behavioral: Waterpipe smoking cessation — The main objective of this study is to compare two levels of intensity of a behavioral intervention for waterpipe smoking cessation, using a randomized controlled trial design. In this trial, brief motivational intervention with self-help materials will be compared with intensive behavioral counseling with four sessions, in order to test the efficacy of each of these interventions. This pilot testing will help us; 1) test the potential efficacy of the developed intervention, 2) fine-tune the intervention in terms of content and format, and 3) assess issues related to recruitment and retention. Thus, feedback from participants and intervention staff will form an essential part of this pilot study to assess the adopted approaches and suggest appropriate modifications.

SUMMARY:
The study is a two-group parallel arm randomized clinical trial, to be conducted at the Syrian Center for Tobacco Studies (SCTS) in Aleppo, Syria.

DETAILED DESCRIPTION:
The study is a two-group parallel arm randomized clinical trial, to be conducted at the Syrian Center for Tobacco Studies (SCTS) in Aleppo, Syria. Subjects will be recruited by flyers, ads, and word of mouth. Smokers who are interested in receiving free stop-smoking assistance as part of a research study will be asked to contact the study office at the SCTS.

Eligibility will be determined by a brief phone screen to determine age, number of years as a smoker and current amount smoked per week, and medical history. Individuals who meet these requirements will be invited to an orientation/screening session at the SCTS to learn more about the study. At the orientation/screening session, the study will be described to interested individuals, their questions will be answered, and those interested in participating will be asked to sign the informed consent document. Participants then will provide baseline demographic information (age, gender, ethnicity, residence, marital status, education, occupation, income) and smoking related information (smoking history, level of dependence, interest in quitting, medical history), and answer other study questionnaires (e.g., self-efficacy, stages of change, and withdrawal symptoms, depression or mood scale). Body weight will be assessed with a calibrated balance-beam scale.

Participants will then be randomized to one of two intervention groups. Subjects in arm A will receive a brief (approximately 15 minute) motivational and educational intervention, delivered by a trained physician from the SCTS, plus written self-help materials. The self-help materials will be adapted and translated into Arabic from existing validated materials from the American Cancer Society and the University of Memphis School of Public Health.

Subjects in Arm B will receive behavioral counseling intervention conducted by a trained physician at the SCTS cessation clinic. Both self-help materials and behavioral intervention will be adapted from established clinical practice guidelines for cigarette smokers (Fiore et al., 2008), experience gained at SCTS with cigarette smokers, and information about the waterpipe gained from previous epidemiological, ethnographic, and clinical studies conducted by the SCTS. Subjects will be requested to do "homework" before the session to facilitate this process. Subjects will be asked to identify high-risk situations and difficulties in previous cessation attempts and will be walked through a series of suggestions in the event of a slip. We also will provide 3 brief (approximately 10 minute) phone calls to subjects during the 90 day follow-up period. These calls are used to identify early relapse, encourage participants, and provide support. In addition, they are used to review materials and information provided during the sessions.

All subjects (Arms A and B) will undergo follow-up assessment at 3 months post-cessation. Data collected at the 3-month follow-up will include expired air carbon monoxide level and several self-report measures, including smoking status, stage of change, and depressive symptomatology. In addition, subjects will be administered a semi-structured questionnaire to assess the perceived usefulness and appropriateness of several features of the cessation intervention (e.g., helpfulness of the interventionist and self-help materials, convenience of the timing and location of the sessions, and usefulness of the phone calls), along with suggestions for improving the intervention. All subjects will receive reminder phone call before the follow-up visits.

All intervention providers will undergo six hours of training for smoking cessation intervention counseling. This training will include general training on intervention delivery, based on current clinical practice standards in developed countries and specific training on study protocols using standardized intervention training materials developed at the University of Memphis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-60 years)
* regular water pipe smokers in Aleppo(at least twice per week for past year)
* interested in quitting
* access to a telephone

Exclusion Criteria:

* unstable cardiovascular, psychiatric, or other debilitating diseases
* inability to provide informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 3 months post-cessation
  The endpoint of cessation will be defined as no self-reported tobacco use, confirmed by expired carbon monoxide of less than 10ppm, at the 3 month post-cessation follow-up visit. Three indicators of cessation will be assessed, including prolonged abstinence (no smoking after two weeks post-quit date), continuous abstinence (no smoking after the quit date), and point-prevalent abstinence (no smoking for the past 7 days).

SECONDARY OUTCOMES:
Stage of change | 3 months post-cessation
  Stage of change in the cessation process (pre-contemplation, contemplation, preparation, action, relapse) based on Prochaska & DiClemente's transtheoretical model.
Depressive symptomatology | 3 months post-cessation
  Self-reported symptoms of depression, based on the CES-D
Intervention acceptability | 3 months post-cessation
  Self-report process measures will be used to assess subject perceptions of helpfulness of the interventionist and self-help materials, convenience of the timing and location of intervention sessions, and usefulness of brief phone intervention contacts.
Fagerström Test for Nicotine Dependence (FTND) | 3 months post-cessation
  To assess smokers'degree of nicotine dependence. Based on Heatherton TF et al. The Fagerström Test for Nicotine Dependence: a revision of the Fagerström Tolerance Questionnaire. Br J Addict. 1991;86:1119-1127.
Social Support | 3 months post-cessation
  To assess smokers'perceived social support. Based on Procidano ME & Heller K. Measures of perceived social support from friends and from family: three validation studies. Am J Community Psychol. 1983;11:1-24.
Smoking-specific self-efficacy | 3 months post-cessation
  To assess smokers' confidence in his/her ability to keep from smoking in a range of different situations. Based on Velicer WF et al. Relapse situations and self-efficacy: an integrative model. Addict Behav. 1990;15:271-283.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D. Ward, PhD, Principal Investigator — The University of Memphis and The Syrian Center for Tobacco Studies
Locations (1):
- Syrian Center for Tobacco Studies, Aleppo, Syria